CLINICAL TRIAL: NCT00859469
Title: Oxaliplatin (Eloxatin®) Plus Gemcitabine as First or Second-line Chemotherapy for Patients With Malignant Pleural or Peritoneal Mesothelioma: A Phase II Clinical Trial
Brief Title: Eloxatin® Plus Gemcitabine Chemotherapy for Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAA2861
Record Dates: First submitted 2009-03-09; First posted 2009-03-11 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Mesothelioma
Keywords: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Oxaliplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxaliplatin and Gemcitabine (Experimental): Gemcitabine 1000 mg/m² IV infusion over 90 minutes, then Oxaliplatin 100 mg/m² IV infusion over 2 hours repeated for 14 days up to 6 cycles
  Interventions: Drug: Oxaliplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin 100 mg/m2 IV infusion for 2 hours
  Other Names: Eloxatin
Drug: Gemcitabine — Gemcitabine 1000mg/m2 IV infusion for 90 minutes
  Other Names: Gemzar

SUMMARY:
In patients with pleural or peritoneal mesothelioma, what is the response rate to combined Oxaliplatin (ELOXATIN®) and Gemcitabine chemotherapy?

DETAILED DESCRIPTION:
Oxaliplatin (ELOXATIN®) is an organoplatinum complex which exerts its cytotoxic effect chiefly through inhibition of tumoral DNA synthesis and repair, leading to cellular apoptosis. The antiproliferative activity of oxaliplatin has been shown to approximate that of cisplatin or carboplatin in different tumor types.

This is a phase II clinical trial of Oxaliplatin (ELOXATIN®) plus gemcitabine as first or secondline chemotherapy for patients with malignant pleural or peritoneal mesothelioma. This study aims to determine the objective tumor response rate for Oxaliplatin plus gemcitabine given every 14 days in patients with malignant pleural mesothelioma and/or malignant peritoneal mesothelioma who have no more than one prior chemotherapy regimen. A total of 29 patients are expected to be enrolled in the study, each with a participation duration of 6 months.

Patients will be screened using standard health care assessments and tests. All of these tests must be done within 4 weeks before patients begin treatment. Patients who are deemed eligible will start the treatment cycle, defined as an interval of 14 days, and comprising of treatment with Gemcitabine followed immediately by Oxaliplatin. The study drugs will be administered in the following manner: Gemcitabine, at 1000 mg/m² IV infusion over 90 minutes, then Oxaliplatin, at 100 mg/m² IV infusion over 2 hours.

In the absence of specific indications for discontinuation of study drugs, patients will routinely be offered 6 cycles of therapy. Further cycles may be given if in the opinion of the investigator this is in the patient's best interest.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignant pleural or peritoneal mesothelioma epithelial, sarcomatoid, or mixed subtype, not amenable to curative treatment with surgery. Patients with pleural mesothelioma will be clinically staged using the International Mesothelioma Interest Group staging criteria. Note that there is no staging system for peritoneal mesothelioma and those patients will only be followed for survival. Patients may be entered based on local pathology.
* Disease status must be that of measurable disease as defined by modified Southwest Oncology Group (SWOG) criteria.

  * Measurable disease: The presence of at least one measurable lesion. If only one lesion is present, the neoplastic nature of the disease site should be confirmed by histology.
  * Measurable lesions: Lesions that can be accurately measured in at least one dimension with the longest diameter ≥20 mm using conventional techniques or ≥10 mm using spiral computerized tomography (CT) scans. At least one level must have one rind measurement ≥15 mm.
* CT (specifically spiral CT) scans and magnetic resonance imaging (MRI) are the preferred methods of measurement.
* Clinically detected lesions will only be considered measurable when they are superficial (e.g., skin nodules and palpable lymph nodes).
* For the case of skin lesions, documentation by color photography, including a ruler to estimate the size of the lesion is required.

NOTE: Neither pleural effusions nor positive bone scans are considered measurable.

* Patients may have undergone pleurodesis. If pleurodesis was performed, there must be at least a 2-week delay before Oxaliplatin or gemcitabine is administered. If the original CT scan occurred prior to the pleurodesis, an additional CT scan is required 2 weeks or longer after the pleurodesis, which will then be considered the baseline scan.

NOTE: For patients with clinically significant pleural effusions or ascites, consideration should be given to draining the fluid.

* Performance status of 0, 1 or 2 on Eastern Cooperative Oncology Group (ECOG) Performance Status Scale (after any palliative measures including pleural drainage have occurred).
* Estimated life expectancy of at least 12 weeks.

Exclusion Criteria:

* More than one previous regimen of systemic chemotherapy. Prior intracavitary cytotoxic drugs will count as a prior regimen, unless given for the purpose of pleurodesis. Immunomodulators will not be regarded as chemotherapy. Prior systemic treatment with pemetrexed plus a platinum compound will not be a contraindication for gemcitabine-oxaliplatin.
* Prior radiation therapy to the target lesion, unless the lesion is clearly progressing and the interval between the most recent radiation therapy and enrollment is at least 4 weeks.
* Active infection (at the discretion of the investigator).
* Pregnancy or breast feeding.
* Serious concomitant systemic disorders (including oncologic emergencies) incompatible with the study (at the discretion of the investigator).
* Patients with a "currently active" second malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix are not to be registered. Patients who are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse.
* Use of any investigational agent within 4 weeks before enrollment into the study.
* Disease which cannot be radiologically imaged.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-04; Primary Completion 2009-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert N Taub, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will be screened using standard health care assessments and tests. All of these tests must be done within 4 weeks before patients begin treatment.
Pre-assignment Details: Patients who are deemed eligible will start the treatment cycle, defined as an interval of 14 days, and comprising of treatment with Gemcitabine followed immediately by Oxaliplatin.
Groups:
- Oxaliplatin and Gemcitabine: The study drugs will be administered in the following manner: Gemcitabine, at 1000 mg/m² IV infusion over 90 minutes, then Oxaliplatin, at 100 mg/m² IV infusion over 2 hours.
Period: Overall Study
Arm/Group | Oxaliplatin and Gemcitabine
Started | 29
6 Cycles | 16
Completed | 1
Not Completed | 28
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 9
Not completed — Withdrawal by Subject | 1
Not completed — Death | 16

BASELINE CHARACTERISTICS:
Arm/Group | Oxaliplatin and Gemcitabine
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 29
Primary Site [Number; unit: participants] — Pleural vs. Peritoneal
  participants
    Pleural | 16
    Peritoneal | 13
Pathologic Subtype [Number; unit: participants] — Epithelioid vs. Sarcomatoid vs. Biphasic
  participants
    Epithelioid | 19
    Sarcomatoid | 3
    Biphasic | 7
Prior chemotherapy regimens [Number; unit: participants]
  0 | 11
  1 or more | 18

OUTCOME MEASURES:

1. Primary Outcome: Best Response
Description: Radiologic response by RECIST criteria will be compared between baseline and at 2 months. Disease assessment: Two objective status determinations of CR before progression are required for a best response of CR. Two determinations of PR or better before progression, but not qualifying for a CR, are required for a best response of PR. Two determinations of stable/no response or better before progression, but not qualifying as CR or PR are required for a best response of stable/no response.
Time Frame: Two months
Population: intention to treat principle
Measure: Number; unit: participants
Arm/Group | Oxaliplatin and Gemcitabine
Number analyzed (Participants) | 29
participants
  Complete Response | 0
  Partial Response | 7
  Stable Disease | 11
  Progressive Disease | 11

2. Secondary Outcome: Overall Survival
Time Frame: 50 months
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oxaliplatin and Gemcitabine
Number analyzed (Participants) | 29
months | 8 [4 to 14]

3. Secondary Outcome: Progression-free Survival
Description: Time to radiologic disease progression or death
Time Frame: 50 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oxaliplatin and Gemcitabine
Number analyzed (Participants) | 29
months | 5 [2 to 7]

ADVERSE EVENTS:
Time Frame: 50 months
Arm/Group | Oxaliplatin and Gemcitabine
Serious Adverse Events (participants affected / at risk) | 11/28
Other Adverse Events (participants affected / at risk) | 27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin and Gemcitabine (N=28)
Anemia (Blood and lymphatic system disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Elevated alkaline phosphatase (Hepatobiliary disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 3
Elevated AST (Hepatobiliary disorders) | 3
Elevated ALT (Hepatobiliary disorders) | 3
Elevated Bilirubin (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Oxaliplatin and Gemcitabine
Leukopenia (Blood and lymphatic system disorders) | 5/26
Thrombocytopenia (Blood and lymphatic system disorders) | 16/28
Anemia (Blood and lymphatic system disorders) | 23/26
Elevated alkaline phosphatase (Hepatobiliary disorders) | 15/26
Elevated AST (Hepatobiliary disorders) | 13/26
Elevated ALT (Hepatobiliary disorders) | 14/26
Nausea/Vomiting (Gastrointestinal disorders) | 9/29
Diarrhea (Gastrointestinal disorders) | 2/29
Peripheral neuropathy (Nervous system disorders) | 11/29
Fever (General disorders) | 2/29
Alopecia (Skin and subcutaneous tissue disorders) | 2/29
Vertigo (Nervous system disorders) | 2/29
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes